CLINICAL TRIAL: NCT01019278
Title: A Feasibility and Phase II Study of Proton Beam Radiotherapy for Patients With Cervical Cancer and FDG-PET Positive Para-aortic Lymph Nodes
Brief Title: Proton Beam Radiation Therapy and Cisplatin in Treating Patients With Stage IB, Stage II, Stage III, or Stage IVA Cervical Cancer and Positive Lymph Nodes
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 22808; NCI-2009-01350
Record Dates: First submitted 2009-11-18; First posted 2009-11-24 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2016-09

CONDITIONS: Cervical Cancer; Stage IB Cervical Cancer; Stage IIA Cervical Cancer; Stage IIB Cervical Cancer; Stage III Cervical Cancer; Stage IVA Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Proton Therapy; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm I (Experimental): Patients undergo external proton beam radiotherapy once daily, 5 times per week, for up to 9 weeks. Patients also receive cisplatin IV once weekly for 6 weeks during radiotherapy.
  Interventions: Radiation: proton beam radiation therapy; Radiation: radiation therapy treatment planning/simulation; Drug: cisplatin

INTERVENTIONS:
Radiation: proton beam radiation therapy — Undergo external proton beam radiation
Radiation: radiation therapy treatment planning/simulation
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP; Neoplatin; PDD

SUMMARY:
RATIONALE: Specialized radiation therapy, such as proton beam radiotherapy, that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving radiation therapy with chemotherapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving proton beam radiation therapy together with cisplatin works in treating patients with stage IB, stage II, stage III, or stage IVA cervical cancer and positive lymph nodes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of proton beam radiotherapy in patients with cervical cancer and FDG-positive para-aortic lymph nodes.

SECONDARY OBJECTIVES:

I. To determine the incidence of acute toxicity of concurrent weekly cisplatin chemotherapy in addition to pelvic and para-aortic irradiation using proton radiotherapy with intracavitary brachytherapy in patients with carcinoma of the uterine cervix with pelvic and para-aortic nodal involvement as demonstrated by FDG-PET.

II. To assess late complications from irradiation using proton beam therapy in place of conventional photon beam therapy.

III. To compare the dose distribution to tumor and surrounding normal structures using DVHs (Dose Volume Histograms) generated from the proton plan used to treat the patient and the photon plan generated for comparison purposes.

IV. To evaluate whether there is a benefit to concurrent weekly cisplatin chemotherapy in addition to pelvic and para-aortic proton beam radiotherapy with intracavitary brachytherapy as evidenced by time to local failure, time to distant failure, time to other failures and overall survival in patients with carcinoma of the uterine cervix with pelvic and para-aortic nodal involvement as demonstrated by FDG-PET.

OUTLINE:

Patients undergo CT, MRI, or FDG-PET imaging scans for radiotherapy treatment planning. Patients then undergo external proton beam radiotherapy once daily, 5 times per week, for up to 9 weeks. Patients also receive cisplatin IV once weekly for 6 weeks during radiotherapy. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years and then annually for 3 years.

ELIGIBILITY:
Inclusion

* Patients must have histologically documented carcinoma of the uterine cervix
* FIGO Stage IB to IVA
* Patients must have no distant metastases apart from positive lymph nodes by FDG PET
* Patients must have a Karnofsky Performance Status of >= 60
* Treatment plan includes cisplatin and patient has no medical contraindications to the administration of cisplatin
* Adequate bone marrow function: WBC >= 3000/mm^3; platelets >= 75,000 mm^3
* Adequate renal function: creatinine =< 2.0 mg/dl (urinary diversion is permitted to improve renal function)
* Patients must have bilirubin =< 1.5 mg/dl
* Ability to understand and the willingness to sign a written informed consent document

Exclusion

* FDG PET Scan evidence of distant disease
* No prior surgery for treatment of disease other than exploratory laparotomy or biopsy will be allowed
* No previous systemic chemotherapy will be allowed
* No prior pelvic radiation therapy is permitted other than transvaginal irradiation to control bleeding will be allowed
* Women of childbearing potential who have a positive result on screening serum pregnancy test

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08-18

PRIMARY OUTCOMES:
Feasibility
Acute toxicity, as assessed by NCI CTC Version 4.0 | Within 60-90 days following completion of proton therapy

SECONDARY OUTCOMES:
Late toxicity, as assessed by RTOG/EORTC late morbidity scoring system | More than 90 days after starting therapy
Clinical efficacy (time to local failure, time to distant failure, overall survival)

CONTACTS AND LOCATIONS:
Overall Officials: Lillie Lin, Principal Investigator — Abramson Cancer Center at Penn Medicine